CLINICAL TRIAL: NCT06088784
Title: A Randomized, Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics of Single and Multiple Doses as Well as the Food Effect of Orally Administered ATH-399A in Healthy Adult Participants
Brief Title: A Study Assessing the Safety of Oral ATH-399A in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HanAll BioPharma Co., Ltd. (Industry)
Collaborators: NurrOn Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HL192-PD-CA-P101; 230119 (Other: Syneos Health)
Record Dates: First submitted 2023-10-05; First posted 2023-10-18 (Actual); Results first posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers
Keywords: ATH399A; HL192; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Parts 1a and 2 are double-blind and Part 1b is open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- Part 1a (Single Ascending Doses (SAD)): ATH-399A (Experimental): Participants will receive single oral dose of ATH-399A capsule at 5mg, 10mg, 20mg, 40mg, 80mg.
  Interventions: Drug: ATH-399A
- Part 1a (SAD): Placebo (Placebo Comparator): Participants will receive single oral dose of placebo-matched to ATH-399A capsule.
  Interventions: Drug: Placebo
- Part 1b (High calorie): ATH-399A (Experimental): Participants will receive single oral dose of ATH-399A capsule after high-calorie, high-fat breakfast and then will cross over to receive single oral dose of ATH-399A capsule after fasting.
  Interventions: Drug: ATH-399A
- Part 1b (Fasting): ATH-399A (Experimental): Participants will receive single oral dose of ATH-399A capsule after fasting and then will cross over to receive single oral dose of ATH-399A capsule after high-calorie, high-fat breakfast.
  Interventions: Drug: ATH-399A
- Part 2 (Multiple Ascending doses (MAD)): ATH-399A (Experimental): Participants will receive once daily (QD) dose of ATH-399A capsules from Day 1 to Day 12 in fasted state.
  Interventions: Drug: ATH-399A
- Part 2 (MAD): Placebo (Placebo Comparator): Participants will receive QD dose of placebo-matched to ATH-399A capsules from Day 1 to Day 12 in fasted state.
  Interventions: Drug: Placebo
- Additional Cohort (Ages 56-80 years old): ATH-399A (Experimental): Participants will receive QD dose of ATH-399A capsules from Day 1 to Day 12 in fasted state following MAD dosing.
  Interventions: Drug: ATH-399A
- Additional Cohort: (Ages 56-80 years old) Placebo (Placebo Comparator): Participants will receive QD dose of placebo-matched to ATH-399A capsules from Day 1 to Day 12 in fasted state following MAD dosing.
  Interventions: Drug: Placebo
- Part 1a - ATH-399A 20 mg (Experimental): Participants will receive single oral dose of 20mg of ATH-399A capsule
  Interventions: Drug: 20mg ATH-399A capsule
- Part 1a (Single Ascending Doses (SAD)): ATH-399A 10 mg (Experimental): Participants will receive single oral dose of 10mg of ATH-399A capsule
  Interventions: Drug: ATH-399A 10 mg
- Part 1a (Single Ascending Doses (SAD)): ATH-399A 5 mg (Experimental): Participants will receive single oral dose of 5mg of ATH-399A capsule
  Interventions: Drug: 5 mg ATH-399A capsule
- Part 1a (Single Ascending Doses (SAD)): ATH-399A 40 mg (Experimental): Participants will receive single oral dose of 40mg of ATH-399A capsule
  Interventions: Drug: 40mg ATH-399A capsule
- Part 1a (Single Ascending Doses (SAD)): ATH-399A 80 mg (Experimental): Participants will receive single oral dose of 80mg of ATH-399A capsule
  Interventions: Drug: 80mg ATH-399A capsule

INTERVENTIONS:
Drug: ATH-399A — Orally administered drug in capsule form.
  Other Names: ATH-399A, HL192
  Arms: Additional Cohort (Ages 56-80 years old): ATH-399A; Part 1a (Single Ascending Doses (SAD)): ATH-399A; Part 1b (Fasting): ATH-399A; Part 1b (High calorie): ATH-399A; Part 2 (Multiple Ascending doses (MAD)): ATH-399A
Drug: Placebo — Orally administered drug in capsule form.
  Arms: Additional Cohort: (Ages 56-80 years old) Placebo; Part 1a (SAD): Placebo; Part 2 (MAD): Placebo
Drug: ATH-399A 10 mg — Participants will receive single oral dose of 10 mg of ATH-399A capsule
  Arms: Part 1a (Single Ascending Doses (SAD)): ATH-399A 10 mg
Drug: 5 mg ATH-399A capsule — Participants will receive single oral dose of 5mg of ATH-399A capsule
  Arms: Part 1a (Single Ascending Doses (SAD)): ATH-399A 5 mg
Drug: 20mg ATH-399A capsule — Participants will receive single oral dose of 20mg of ATH-399A capsule
  Arms: Part 1a - ATH-399A 20 mg
Drug: 40mg ATH-399A capsule — Participants will receive single oral dose of 40mg of ATH-399A capsule
  Arms: Part 1a (Single Ascending Doses (SAD)): ATH-399A 40 mg
Drug: 80mg ATH-399A capsule — Participants will receive single oral dose of 80mg of ATH-399A capsule
  Arms: Part 1a (Single Ascending Doses (SAD)): ATH-399A 80 mg

SUMMARY:
This study will evaluate the safety, tolerability and pharmacokinetics of single and multiple doses of ATH-399A in healthy adults and also evaluate the effect of food on ATH-399A in order to develop mechanism-based and/or disease-modifying treatments for Parkinson Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, as determined by the Investigator based on a medical evaluation including medical history, physical examination, neurological examination, laboratory tests, and cardiac monitoring.
2. Population

   1. Part 1a and 1b: Men and women, age 18-55 years inclusive at the date of screening.
   2. Part 2: Men and women aged 18-55 years inclusive at the date of screening. Additional cohort: Participants of the additional cohort will be of approximately equal numbers of male and post-menopausal or surgically sterile females, with a minimum of 2 of each gender, aged >55-80 years, inclusive.
3. Women of childbearing potential (WOCBP) must be non-pregnant and non-lactating.
4. Postmenopausal women must have had ≥12 months of spontaneous amenorrhea (with follicle-stimulating hormone [FSH] ≥40 milli-international units per milliliter (mIU/mL)).
5. Surgically sterile women are defined as those who have had a hysterectomy and/or bilateral oophorectomy. Women who are surgically sterile must provide verbal confirmation.
6. Male participants who are sexually active with WOCBP must:

   1. Agree to use condoms to protect their partners from becoming pregnant during the study (including washout periods) and not to donate sperm for at least 90 days after the last dose of the study drug, and
   2. Agree to ensure that they and their partners are routinely using a medically approved contraceptive method. It is important that male participants not impregnate others while in the study.
7. Body weight ≥50.0 kilograms (kg) for men and ≥45.0 kg for women and body mass index within the range of 18.0-30.0 kilogram/square meter (kg/m^2) (inclusive).
8. Participants participating in Part 1b must be willing and able to consume the entire high-fat, high-calorie breakfast in the designated timeframe.
9. Participants must understand the nature of the study, must be willing to participate in the study, and must provide signed and dated written informed consent in accordance with local regulations before the conduct of any study-related procedures.
10. Participants must be, in the opinion of the Investigator, able to participate in all scheduled evaluations, likely to complete all required tests, and likely to be compliant.
11. Participants must be fluent in English or French.
12. Participants must agree not to post any personal medical data related to the study or information related to the study on any website or social media site.

Exclusion Criteria:

1. A positive urine cotinine, drug screen, or alcohol breath test at screening or Day -1.
2. Any history of psychiatric disorders, including substance use disorders, according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria that requires current treatment with psychiatric medications. Participants with mild anxiety or depression which is stable for >6 months are permitted.
3. History of drug abuse within 1 year prior to screening or recreational use of soft drugs (such as marijuana) within 1 month or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within 3 months prior to screening.
4. A diagnosis of intellectual disability (intellectual developmental disorder) or mental retardation.
5. A serious mental illness, dementia, or other neuropsychiatric disorder that would interfere with participation in the trial, or ability to provide informed consent in the opinion of the Investigator.
6. Any active suicidal ideation as indicated by the C-SSRS (score of ≥4) or history of suicidal behavior within the 12 months prior to screening.
7. A positive Hepatitis B surface antigen or positive Hepatitis C antibody result at screening.
8. A positive test at screening for human immunodeficiency virus (HIV) antigen or antibody or a history of positive test.
9. Alanine aminotransferase or aspartate aminotransferase levels greater than 1.2 times the ULN at screening or Day -1.
10. Frequently use (>5 per week) any tobacco-containing (e.g., cigar, cigarette or snuff) or nicotine-containing product (e.g., nicotine chewing gum, nicotine plasters, or other product used for smoking cessation) within 30 days prior to the first dose administration. Use of any tobacco- or nicotine-containing product is prohibited within 2 weeks of first dose administration through completion of the in-clinic stay for the SAD (Parts 1a and 1b) and until after the final study visit for the MAD (Part 2).
11. History of alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to screening that exceeds 10 units for women or 15 units for men of alcohol per week (1 unit = 340 mL of beer 5%, 140 mL of wine 12%, or 45 mL of distilled alcohol 40%).
12. Regularly consumed (e.g., more days than not) excessive quantities of xanthine-containing beverages (e.g., more than 2 cups of coffee or the equivalent per day) within 1 week prior to screening or between screening and first dose administration, or unwillingness to refrain from xanthine-containing beverages during the in-clinic stay.
13. Received or used an investigational product (including placebo) or device within the following time period prior to the first dosing day in the current study: 30 days or 5 half-lives (whichever is longer). For biological products, administration of a biological product within 90 days prior to the first dosing, or concomitant participation in an investigational study involving no drug or device administration.
14. Other than those medications outlined in the protocol body and those allowed in the MAD additional cohort, use of prescription or non-prescription drugs, herbal, and dietary supplements (including St John's Wort) within 7 days (or 28 days if the drug is a potential hepatic enzyme inducer) or 5 half-lives (whichever is longer) prior to first dose administration, unless in the opinion of the Investigator and Medical Monitor, the medication will not interfere with the study procedures or compromise participant safety.
15. History of clinically significant sensitivity to any of the study drugs, or components thereof, or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates their participation.
16. Donation of plasma within 7 days prior to the first dosing or donation or loss of 500 mL or more of whole blood within 8 weeks prior to the first dosing.
17. A positive pregnancy test or lactation.
18. A history or presence of any disease, condition, or surgery likely to affect drug absorption, distribution, metabolism, or excretion. Participants with a history of cholecystectomy should be excluded.
19. A history or presence of a clinically significant hepatic, renal, gastrointestinal, cardiovascular, endocrine, pulmonary, ophthalmologic, immunologic, hematologic, dermatologic, or neurologic abnormality. Participants with fully resolved childhood asthma with no hospitalizations or recurrence in adulthood are permitted to enroll. For the additional cohort in Part 2, any of the above is acceptable where the condition is stable for >6 months and, in the opinion of the Investigator, it does not impact participant safety.
20. A clinically significant abnormality on physical examination, neurological examination, electrocardiogram (ECG), or laboratory evaluations at screening and Day -1.
21. A QT interval measurement corrected according to the Fridericia rule (QTcF) > 450 milliseconds (msec) during controlled rest at screening and Day -1, or family history of long QT syndrome.
22. Any clinically significant abnormalities in rhythm, conduction, or morphology of the resting ECG and any abnormalities in the 12-lead ECG that, in the judgment of the Investigator or Medical Monitor, may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology or left ventricular hypertrophy.
23. A clinically significant vital sign abnormality at screening or between screening and first dose administration.
24. Significant (> 10%) weight loss or gain within 30 days prior to screening or between screening and first dose administration.
25. A history of seizures. The occurrence of a single febrile seizure is not exclusionary.
26. A history of head trauma, including closed head injury with loss of consciousness. Concussions which did not lead to hospitalization or loss of consciousness, and for which there are no ongoing issues, are not exclusionary.
27. A history of symptomatic orthostatic hypotension (i.e., postural syncope).
28. A history of neuroleptic malignant syndrome.
29. A history of chronic urinary tract infections (≥2 times per year).
30. The participant is, in the opinion of the Investigator or Medical Monitor, unlikely to comply with the protocol or is unsuitable for any reason.
31. Currently employed by NurrOn Pharmaceuticals, Inc., HanAll Biopharma Co. Ltd., or HanAll Pharmaceutical Inc., or by a clinical trial site participating in this study, or a first-degree relative of a NurrOn Pharmaceuticals, Inc. or HanAll Pharmaceutical Inc., or HanAll Biopharma Co. Ltd. employee or of an employee at a participating clinical trial site.
32. Unsatisfactory venous access.
33. Unable to swallow oral capsules.
34. Positive result to a coronavirus disease (COVID-19) Polymerase chain reaction (PCR) test.
35. COVID-19 or flu vaccination within 30 days prior to study drug administration or any other vaccination that is judged by the investigator to potentially affect eligibility.
36. Presence of fever (body temperature >37.5°C) (e.g., a fever associated with a symptomatic viral or bacterial infection) within 2 weeks prior to the first dosing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-04-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Syneos Quebec Canada, Québec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part 1a: 40 participants randomized Part 1b: 12 participants randomized Part 2: 24 participants randomized
Groups:
- Part 1a (SAD): ATH-399A 5 mg: Each participant received a single oral dose of 5 mg of ATH-399A.
- Part 1a (SAD): ATH-399A 10 mg: Each participant received a single oral dose of 10 mg of ATH-399A.
- Part 1a (SAD): ATH-399A 20 mg: Each participant received a single oral dose of 20 mg of ATH-399A.
- Part 1a (SAD): ATH-399A 40 mg: Each participant received a single oral dose of 40 mg of ATH-399A.
- Part 1a (SAD): ATH-399A 80 mg: Each participant received a single oral dose of 80 mg of ATH-399A.
- Part 1a (SAD): Placebo; Part 2 (MAD): Placebo: Each participant received a single dose of matching placebo.
- Part 1b (Food Effect): ATH-399A 40 mg, Sequence AB; Part 1b (Food Effect): ATH-399A 40 mg, Sequence BA: Participants in Part 1b were randomized to one of the 2 arms to receive study drugs in the cross-over sequence AB or BA.
  * Treatment A: ATH-399A 40 mg was administered following a high-fat, high-calorie meal.
  * Treatment B: Participants were restricted from eating 10 hours prior to and 4 hours following ATH-399A 40 mg administration.
- Part 2 (MAD): ATH-399A 20 mg: Each participant received ATH-399A 20 mg once daily from Day 1 to Day 12. Participants underwent a supervised fast for at least 10 hours prior to dosing, followed by an additional 4 hours of fasting post-dose.
- Part 2 (MAD): ATH-399A 40 mg: Each participant received ATH-399A 40 mg once daily from Day 1 to Day 12. Participants underwent a supervised fast for at least 10 hours prior to dosing, followed by an additional 4 hours of fasting post-dose.
- Part 2 (MAD): ATH-399A 40 mg, Older: Each participant aged >55-80 years received ATH-399A 40 mg once daily from Day 1 to Day 12. Participants underwent a supervised fast for at least 10 hours prior to dosing, followed by an additional 4 hours of fasting post-dose.
Period: Overall Study
Arm/Group | Part 1a (SAD): ATH-399A 5 mg | Part 1a (SAD): ATH-399A 10 mg | Part 1a (SAD): ATH-399A 20 mg | Part 1a (SAD): ATH-399A 40 mg | Part 1a (SAD): ATH-399A 80 mg | Part 1a (SAD): Placebo | Part 1b (Food Effect): ATH-399A 40 mg, Sequence AB | Part 1b (Food Effect): ATH-399A 40 mg, Sequence BA | Part 2 (MAD): ATH-399A 20 mg | Part 2 (MAD): ATH-399A 40 mg | Part 2 (MAD): ATH-399A 40 mg, Older | Part 2 (MAD): Placebo
Started | 6 | 6 | 6 | 6 | 6 | 10 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6 | 6 | 10 | 2 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Exclusion criterion: QTcF >450 msec | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1a (SAD): ATH-399A 5 mg | Part 1a (SAD): ATH-399A 10 mg | Part 1a (SAD): ATH-399A 20 mg | Part 1a (SAD): ATH-399A 40 mg | Part 1a (SAD): ATH-399A 80 mg | Part 1a (SAD): Placebo | Part 1b (Food Effect): ATH-399A 40 mg, Sequence AB | Part 1b (Food Effect): ATH-399A 40 mg, Sequence BA | Part 2 (MAD): ATH-399A 20 mg | Part 2 (MAD): ATH-399A 40 mg | Part 2 (MAD): ATH-399A 40 mg, Older | Part 2 (MAD): Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 6 | 6 | 6 | 6 | 6 | 6 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (8.07) | 35.5 (10.80) | 50.0 (5.29) | 39.0 (8.88) | 42.8 (5.46) | 39.2 (8.88) | 37.0 (13.34) | 41.5 (10.05) | 35.7 (11.72) | 47.0 (6.96) | 64.8 (5.31) | 50.2 (12.64) | 43.07 (11.8292)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 4 | 0 | 4 | 6 | 2 | 3 | 2 | 1 | 3 | 2 | 32
  Male | 3 | 4 | 2 | 6 | 2 | 4 | 4 | 3 | 4 | 5 | 3 | 4 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 2 | 2 | 0 | 3 | 2 | 0 | 3 | 1 | 2 | 19
  Not Hispanic or Latino | 5 | 5 | 4 | 4 | 4 | 10 | 3 | 4 | 6 | 3 | 5 | 4 | 57
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 7
  White | 5 | 5 | 6 | 3 | 6 | 10 | 6 | 6 | 5 | 5 | 6 | 5 | 68
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 168.67 (8.134) | 171.08 (6.931) | 163.73 (8.188) | 176.57 (9.528) | 168.33 (6.439) | 166.70 (12.541) | 170.92 (8.357) | 167.68 (7.427) | 172.70 (10.050) | 171.83 (7.757) | 170.68 (7.105) | 174.25 (8.802) | 170.08 (8.8719)
Weight [Mean (Standard Deviation); unit: kg] | 70.43 (11.316) | 71.83 (7.689) | 64.52 (11.874) | 79.93 (15.591) | 74.25 (12.798) | 67.15 (9.957) | 76.12 (14.787) | 69.20 (11.516) | 72.87 (15.164) | 79.92 (10.198) | 69.92 (11.940) | 76.10 (12.381) | 72.39 (12.1717)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 24.72 (3.277) | 24.50 (1.971) | 23.97 (3.236) | 25.48 (3.388) | 26.03 (3.027) | 24.16 (2.476) | 25.90 (3.551) | 24.60 (3.529) | 24.22 (3.573) | 26.93 (1.507) | 23.87 (2.889) | 24.93 (2.479) | 24.90 (2.8730)

OUTCOME MEASURES:

1. Primary Outcome: Number of TEAEs
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study drug, whether or not considered related to the study drug.
Time Frame: Continuously during study period from baseline to follow-up visit: Part 1a: Day-1 to Day 8, Part 1b: Day-1 to Day 16; and Part 2: Day -1 to Day 19
Measure: Number; unit: Treatment Emergent Adverse Event
Groups:
- Part 1b (Food Effect): ATH-399A 40 mg, Fed: ATH-399A 40 mg was administered following a high-fat, high-calorie meal.
- Part 1b (Food Effect): ATH-399A 40 mg, Fasted: Participants were restricted from eating 10 hours prior to and 4 hours following ATH-399A 40 mg administration.
Arm/Group | Part 1a (SAD): ATH-399A 5 mg | Part 1a (SAD): ATH-399A 10 mg | Part 1a (SAD): ATH-399A 20 mg | Part 1a (SAD): ATH-399A 40 mg | Part 1a (SAD): ATH-399A 80 mg | Part 1a (SAD): Placebo | Part 1b (Food Effect): ATH-399A 40 mg, Fed | Part 1b (Food Effect): ATH-399A 40 mg, Fasted | Part 2 (MAD): ATH-399A 20 mg | Part 2 (MAD): ATH-399A 40 mg | Part 2 (MAD): ATH-399A 40 mg, Older | Part 2 (MAD): Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 12 | 8 | 6 | 6 | 6 | 6
Treatment Emergent Adverse Event | 4 | 2 | 1 | 3 | 2 | 3 | 3 | 1 | 4 | 2 | 10 | 6

2. Primary Outcome: Participants With at Least 1 TEAE
Description: Participants with at least one AE started or after the time of first study drug administration.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1a (SAD): ATH-399A 5 mg | Part 1a (SAD): ATH-399A 10 mg | Part 1a (SAD): ATH-399A 20 mg | Part 1a (SAD): ATH-399A 40 mg | Part 1a (SAD): ATH-399A 80 mg | Part 1a (SAD): Placebo | Part 1b (Food Effect): ATH-399A 40 mg, Fed | Part 1b (Food Effect): ATH-399A 40 mg, Fasted | Part 2 (MAD): ATH-399A 20 mg | Part 2 (MAD): ATH-399A 40 mg | Part 2 (MAD): ATH-399A 40 mg, Older | Part 2 (MAD): Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 12 | 8 | 6 | 6 | 6 | 6
Participants | 4 | 1 | 1 | 2 | 1 | 2 | 3 | 1 | 3 | 2 | 3 | 2

3. Primary Outcome: Serious TEAEs
Description: An SAE was defined as any untoward medical occurrence that, at any dose, met one or more of the criteria listed: Resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or other situations.
Time Frame: as for outcome 1
Measure: Number; unit: Serious Treatment Emergent Adverse Event
Groups:
- Part 2 (MAD): ATH-399A 40 mg, Older: A total of 24 participants were randomized in Part 2. All 24 participants received at least one dose of the study drug (active or placebo) and comprised the Safety Population. In accordance with the study protocol, all participants who received at least one dose of In this study part, this cohort included older population, aged >55 - 80 years
Arm/Group | Part 1a (SAD): ATH-399A 5 mg | Part 1a (SAD): ATH-399A 10 mg | Part 1a (SAD): ATH-399A 20 mg | Part 1a (SAD): ATH-399A 40 mg | Part 1a (SAD): ATH-399A 80 mg | Part 1a (SAD): Placebo | Part 1b (Food Effect): ATH-399A 40 mg, Fed | Part 1b (Food Effect): ATH-399A 40 mg, Fasted | Part 2 (MAD): ATH-399A 20 mg | Part 2 (MAD): ATH-399A 40 mg | Part 2 (MAD): ATH-399A 40 mg, Older | Part 2 (MAD): Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 12 | 8 | 6 | 6 | 6 | 6
Serious Treatment Emergent Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Suicidal Ideation and/or Behavior Detected in Columbia Suicidality Severity Rating Scale (C-SSRS)
Description: Number of participant whose answers indicate suicidal ideation and/or behavior at follow-up.
Time Frame: Part 1a, 1b: Screening, Day -1, Follow-up (1a - Day 16; 1b - Day 19); Part 2: Screening, Day -1, Day 13 (Discharge or early termination)
Population: Participants in each part were combined for reporting results given there were 0 reports across the study.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1a (SAD) 5 mg: Each participant received a single dose of either 5 mg ATH-399A or matching placebo.
- Part 1b (Food Effect) Fed; Part 1b (Food Effect) Fasted: Participants in Part 1b were randomized to one of the 2 arms to receive study drugs in the cross-over sequence AB or BA.
  * Treatment A: ATH-399A 40 mg was administered following a high-fat, high-calorie meal.
  * Treatment B: Participants were restricted from eating 10 hours prior to and 4 hours following ATH-399A 40 mg administration.
- Part 2 (MAD) 20 mg: Each participant (aged 18-55 yo) received ATH-399A 20 mg once daily from Day 1 to Day 12. Participants underwent a supervised fast for at least 10 hours prior to dosing, followed by an additional 4 hours of fasting post-dose.
- Part 1a (SAD) 10 mg: Each participant received a single dose of either 10 mg ATH-399A or matching placebo.
- Part 1a (SAD) 20 mg: Each participant received a single dose of either 20 mg ATH-399A or matching placebo.
- Part 1a (SAD) 40 mg: Each participant received a single dose of either 40 mg ATH-399A or matching placebo.
- Part 1a (SAD) 80 mg: Each participant received a single dose of either 80 mg ATH-399A or matching placebo.
- Part 1a (SAD) placebo: Each participant received a sing dose of placebo.
- Part 2 (MAD) 40 mg: Each participant (aged 18-55 yo) received ATH-399A 40 mg once daily from Day 1 to Day 12. Participants underwent a supervised fast for at least 10 hours prior to dosing, followed by an additional 4 hours of fasting post-dose.
- Part 2 (MAD) 40 mg Older: Each participant (aged >55 yo) received ATH-399A 40 mg once daily from Day 1 to Day 12. Participants underwent a supervised fast for at least 10 hours prior to dosing, followed by an additional 4 hours of fasting post-dose.
- Part 2 (MAD) placebo: Each participant received ATH-399A pacebo once daily from Day 1 to Day 12. Participants underwent a supervised fast for at least 10 hours prior to dosing, followed by an additional 4 hours of fasting post-dose.
Arm/Group | Part 1a (SAD) 5 mg | Part 1b (Food Effect) Fed | Part 2 (MAD) 20 mg | Part 1a (SAD) 10 mg | Part 1a (SAD) 20 mg | Part 1a (SAD) 40 mg | Part 1a (SAD) 80 mg | Part 1a (SAD) placebo | Part 1b (Food Effect) Fasted | Part 2 (MAD) 40 mg | Part 2 (MAD) 40 mg Older | Part 2 (MAD) placebo
Number analyzed (Participants) | 6 | 12 | 6 | 6 | 6 | 6 | 6 | 10 | 8 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: QTcF Analysis
Description: Participants with abnormal QTcF on ECG (pooled data from the whole study duration)
Time Frame: From baseline to follow up visit: Part 1a: Day-1 to Day 8, Part 1b: Day-1 to Day 16; and Part 2: Day -1 to Day 19
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1a (SAD): ATH-399A 5 mg | Part 1a (SAD): ATH-399A 10 mg | Part 1a (SAD): ATH-399A 20 mg | Part 1a (SAD): ATH-399A 40 mg | Part 1a (SAD): ATH-399A 80 mg | Part 1a (SAD): Placebo | Part 1b (Food Effect): ATH-399A 40 mg, Fed | Part 1b (Food Effect): ATH-399A 40 mg, Fasted | Part 2 (MAD): ATH-399A 20 mg | Part 2 (MAD): ATH-399A 40 mg | Part 2 (MAD): ATH-399A 40 mg, Older | Part 2 (MAD): Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 12 | 8 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 0

6. Primary Outcome: Changes in Diastolic Blood Pressure
Description: Diastolic blood pressure baseline value measured at basline Day 1 pre dose and Day 1 1 hour post dosing
Time Frame: Day 1: predose and 1 hour post dosing
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part 1a (SAD): ATH-399A 5 mg | Part 1a (SAD): ATH-399A 10 mg | Part 1a (SAD): ATH-399A 20 mg | Part 1a (SAD): ATH-399A 40 mg | Part 1a (SAD): ATH-399A 80 mg | Part 1a (SAD): Placebo | Part 1b (Food Effect): ATH-399A 40 mg, Fed | Part 1b (Food Effect): ATH-399A 40 mg, Fasted | Part 2 (MAD): ATH-399A 20 mg | Part 2 (MAD): ATH-399A 40 mg | Part 2 (MAD): ATH-399A 40 mg, Older | Part 2 (MAD): Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 12 | 8 | 6 | 6 | 6 | 6
mmHg
  Baseline | 68.8 (7.73) | 70.8 (4.07) | 75.8 (7.39) | 70.7 (4.32) | 72.5 (7.87) | 71.0 (6.46) | 69.8 (6.12) | 69.0 (4.81) | 72.8 (3.19) | 72.0 (4.00) | 72.3 (1.97) | 71.5 (7.77)
  1 hour post dosing | 67.5 (6.35) | 69.2 (5.27) | 74.3 (6.74) | 71.8 (6.91) | 70.5 (7.18) | 70.7 (5.89) | 66.1 (6.10) | 70.9 (6.13) | 71.8 (5.12) | 70.8 (3.19) | 75.2 (3.19) | 73.0 (9.57)

7. Primary Outcome: Changes in Systolic Blood Pressure
Description: Systolic blood pressure baseline value measured at basline Day 1 pre dose and Day 1 1 hour post dosing
Time Frame: Day 1 predose and 1 hour postdosing
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part 1a (SAD): ATH-399A 5 mg | Part 1a (SAD): ATH-399A 10 mg | Part 1a (SAD): ATH-399A 20 mg | Part 1a (SAD): ATH-399A 40 mg | Part 1a (SAD): ATH-399A 80 mg | Part 1a (SAD): Placebo | Part 1b (Food Effect): ATH-399A 40 mg, Fed | Part 1b (Food Effect): ATH-399A 40 mg, Fasted | Part 2 (MAD): ATH-399A 20 mg | Part 2 (MAD): ATH-399A 40 mg | Part 2 (MAD): ATH-399A 40 mg, Older | Part 2 (MAD): Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 12 | 8 | 6 | 6 | 6 | 6
mmHg
  1 hour post dosing | 105.8 (7.65) | 110.8 (7.36) | 117.0 (12.55) | 113.8 (10.23) | 108.3 (11.04) | 109.5 (9.00) | 119.9 (13.99) | 116.5 (9.34) | 114.7 (9.50) | 113.8 (5.12) | 123.7 (11.43) | 113.5 (9.38)
  baseline | 107.0 (7.21) | 112.0 (4.20) | 119.7 (12.37) | 111.3 (5.24) | 111.8 (9.64) | 111.6 (9.13) | 111.4 (8.05) | 110.1 (7.83) | 114.3 (5.39) | 114.5 (9.97) | 116.3 (8.89) | 112.7 (11.47)

8. Primary Outcome: Heart Rate Value
Description: Heart rate value measured at Day 1, 1 Hour Post-Dose
Time Frame: Day 1, 1 hour post-dose
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Part 1a (SAD): ATH-399A 5 mg | Part 1a (SAD): ATH-399A 10 mg | Part 1a (SAD): ATH-399A 20 mg | Part 1a (SAD): ATH-399A 40 mg | Part 1a (SAD): ATH-399A 80 mg | Part 1a (SAD): Placebo | Part 1b (Food Effect): ATH-399A 40 mg, Fed | Part 1b (Food Effect): ATH-399A 40 mg, Fasted | Part 2 (MAD): ATH-399A 20 mg | Part 2 (MAD): ATH-399A 40 mg | Part 2 (MAD): ATH-399A 40 mg, Older | Part 2 (MAD): Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 12 | 8 | 6 | 6 | 6 | 6
beats/min | 59.7 (10.27) | 58.3 (6.09) | 55.3 (5.16) | 63.0 (10.81) | 59.8 (6.05) | 64.7 (7.29) | 65.3 (8.86) | 60.6 (5.71) | 62.3 (6.22) | 58.7 (8.29) | 63.0 (9.21) | 61.0 (7.46)

9. Primary Outcome: Temperature Value
Description: Temperature value measured at Day 1, 1 Hour Post-Dose
Time Frame: Day 1, 1 Hour Post-Dose
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | Part 1a (SAD): ATH-399A 5 mg | Part 1a (SAD): ATH-399A 10 mg | Part 1a (SAD): ATH-399A 20 mg | Part 1a (SAD): ATH-399A 40 mg | Part 1a (SAD): ATH-399A 80 mg | Part 1a (SAD): Placebo | Part 1b (Food Effect): ATH-399A 40 mg, Fed | Part 1b (Food Effect): ATH-399A 40 mg, Fasted | Part 2 (MAD): ATH-399A 20 mg | Part 2 (MAD): ATH-399A 40 mg | Part 2 (MAD): ATH-399A 40 mg, Older | Part 2 (MAD): Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 12 | 8 | 6 | 6 | 6 | 6
°C | 36.63 (0.103) | 36.67 (0.121) | 36.72 (0.232) | 36.78 (0.147) | 36.73 (0.216) | 36.78 (0.210) | 36.80 (0.160) | 36.73 (0.116) | 36.93 (0.151) | 36.58 (0.117) | 36.63 (0.207) | 36.70 (0.167)

10. Primary Outcome: Respiratory Rate Value
Description: Respiratory rate value measured at Day 1, 1 Hour Post-Dose
Time Frame: Day 1, 1 Hour Post-Dose
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Part 1a (SAD): ATH-399A 5 mg | Part 1a (SAD): ATH-399A 10 mg | Part 1a (SAD): ATH-399A 20 mg | Part 1a (SAD): ATH-399A 40 mg | Part 1a (SAD): ATH-399A 80 mg | Part 1a (SAD): Placebo | Part 1b (Food Effect): ATH-399A 40 mg, Fed | Part 1b (Food Effect): ATH-399A 40 mg, Fasted | Part 2 (MAD): ATH-399A 20 mg | Part 2 (MAD): ATH-399A 40 mg | Part 2 (MAD): ATH-399A 40 mg, Older | Part 2 (MAD): Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 12 | 8 | 6 | 6 | 6 | 6
breaths/min | 14.7 (2.73) | 16.0 (3.58) | 13.7 (1.51) | 13.0 (3.74) | 14.3 (2.34) | 13.0 (3.30) | 15.5 (3.09) | 14.3 (1.98) | 14.7 (1.03) | 15.0 (1.10) | 13.0 (3.52) | 13.3 (2.07)

11. Primary Outcome: Physical Examination and Neurological Examination Abnormalities Analysis
Description: Participants with abnormal findings on physical and neurological examination (pooled data from the whole study)
Time Frame: Part 1a, 1b, 2: Screening, D-1, D3 (Discharge or early termination), Follow-Up: Part 1a: Day 8, Part 1b: Day 16; and Part 2: Day 19
Measure: Number; unit: Participants
Arm/Group | Part 1a (SAD): ATH-399A 5 mg | Part 1a (SAD): ATH-399A 10 mg | Part 1a (SAD): ATH-399A 20 mg | Part 1a (SAD): ATH-399A 40 mg | Part 1a (SAD): ATH-399A 80 mg | Part 1a (SAD): Placebo | Part 1b (Food Effect): ATH-399A 40 mg, Fed | Part 1b (Food Effect): ATH-399A 40 mg, Fasted | Part 2 (MAD): ATH-399A 20 mg | Part 2 (MAD): ATH-399A 40 mg | Part 2 (MAD): ATH-399A 40 mg, Older | Part 2 (MAD): Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 12 | 8 | 6 | 6 | 6 | 6
Participants | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

12. Primary Outcome: 12-Lead Telemetry Abnormalities Analysis
Description: Participants with abnormal findings on 12-lead telemetry (pooled data from the whole study)
Time Frame: Part 1a, 1b: D1, D2, D3; Part 2: D1, D2, D12, D13 (Discharge or early termination)
Measure: Number; unit: Participants
Arm/Group | Part 1a (SAD): ATH-399A 5 mg | Part 1a (SAD): ATH-399A 10 mg | Part 1a (SAD): ATH-399A 20 mg | Part 1a (SAD): ATH-399A 40 mg | Part 1a (SAD): ATH-399A 80 mg | Part 1a (SAD): Placebo | Part 1b (Food Effect): ATH-399A 40 mg, Fed | Part 1b (Food Effect): ATH-399A 40 mg, Fasted | Part 2 (MAD): ATH-399A 20 mg | Part 2 (MAD): ATH-399A 40 mg | Part 2 (MAD): ATH-399A 40 mg, Older | Part 2 (MAD): Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 12 | 8 | 6 | 6 | 6 | 6
Participants | 2 | 1 | 1 | 1 | 2 | 2 | 5 | 2 | 3 | 1 | 4 | 1

13. Secondary Outcome: AUC0-t
Description: Plasma Pharmacokinetic (PK) parameter: Area Under the Concentration-Time Curve from Time Zero Until the Last Observed Concentration (AUC0-t) for Part 1a, Part 1b and Part 2. AUC0-t was calculated based on several PK blood sampling at times provided in the Outcome Measure Time Frame.
Time Frame: Part 1: Day 1 Pre-dose (within 2 hours of dosing) and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 hours. Part 2: Day 12 Pre-dose (within 2 hours of dosing) and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 hours.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 1a (SAD): ATH-399A 5 mg | Part 1a (SAD): ATH-399A 10 mg | Part 1a (SAD): ATH-399A 20 mg | Part 1a (SAD): ATH-399A 40 mg | Part 1a (SAD): ATH-399A 80 mg | Part 1b (Food Effect): ATH-399A 40 mg, Fed | Part 1b (Food Effect): ATH-399A 40 mg, Fasted | Part 2 (MAD): ATH-399A 20 mg | Part 2 (MAD): ATH-399A 40 mg | Part 2 (MAD): ATH-399A 40 mg, Older
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 12 | 8 | 6 | 6 | 6
h*ng/mL | 34.19 (8.34) | 53.71 (30.15) | 168.62 (73.85) | 481.81 (171.08) | 1093.98 (274.05) | 651.13 (179.31) | 569.69 (189.58) | 450.52 (124.54) | 1337.49 (577.26) | 1601.07 (476.59)

14. Secondary Outcome: AUC0-inf
Description: PK parameter: Area Under The Concentration-Time Curve From Time Zero To Infinity (Extrapolated) (AUC0-inf) for Part 1a, Part 1b and Part 2. AUC0-inf was calculated based on several PK blood sampling at times provided in the Outcome Measure Time Frame.
Time Frame: as for outcome 13
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 1a (SAD): ATH-399A 5 mg | Part 1a (SAD): ATH-399A 10 mg | Part 1a (SAD): ATH-399A 20 mg | Part 1a (SAD): ATH-399A 40 mg | Part 1a (SAD): ATH-399A 80 mg | Part 1b (Food Effect): ATH-399A 40 mg, Fed | Part 1b (Food Effect): ATH-399A 40 mg, Fasted | Part 2 (MAD): ATH-399A 20 mg | Part 2 (MAD): ATH-399A 40 mg | Part 2 (MAD): ATH-399A 40 mg, Older
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 12 | 8 | 6 | 5 | 4
h*ng/mL | 45.92 (9.28) | 86.22 (32.59) | 212.02 (95.27) | 522.19 (172.75) | 1200.69 (320.04) | 720.93 (211.31) | 625.05 (209.54) | 485.14 (134.00) | 1454.58 (629.97) | 1782.88 (504.10)

15. Secondary Outcome: Cmax
Description: PK parameter: Maximal Observed Concentration (Cmax) for Part 1a, Part 1b and Part 2. Cmax was calculated based on several PK blood sampling at times provided in the Outcome Measure Time Frame.
Time Frame: Part 1: Day 1 Pre-dose (within 2 hours of dosing) and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 hours. Part 2: Day 1 Pre-dose (within 2 hours of dosing) and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 hours.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1a (SAD): ATH-399A 5 mg | Part 1a (SAD): ATH-399A 10 mg | Part 1a (SAD): ATH-399A 20 mg | Part 1a (SAD): ATH-399A 40 mg | Part 1a (SAD): ATH-399A 80 mg | Part 1b (Food Effect): ATH-399A 40 mg, Fed | Part 1b (Food Effect): ATH-399A 40 mg, Fasted | Part 2 (MAD): ATH-399A 20 mg | Part 2 (MAD): ATH-399A 40 mg | Part 2 (MAD): ATH-399A 40 mg, Older
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 12 | 8 | 6 | 6 | 6
ng/mL | 1.53 (0.55) | 1.93 (1.03) | 9.11 (5.28) | 20.57 (11.95) | 45.40 (14.51) | 22.50 (7.90) | 22.49 (11.58) | 5.32 (2.46) | 14.21 (10.64) | 13.78 (10.23)

16. Secondary Outcome: Tmax
Description: PK parameter: Time When The Maximal Concentration Is Observed (Tmax) for Part 1a, Part 1b and Part 2. Tmax was calculated based on several PK blood sampling at times provided in the Outcome Measure Time Frame.
Time Frame: as for outcome 15
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1a (SAD): ATH-399A 5 mg | Part 1a (SAD): ATH-399A 10 mg | Part 1a (SAD): ATH-399A 20 mg | Part 1a (SAD): ATH-399A 40 mg | Part 1a (SAD): ATH-399A 80 mg | Part 1b (Food Effect): ATH-399A 40 mg, Fed | Part 1b (Food Effect): ATH-399A 40 mg, Fasted | Part 2 (MAD): ATH-399A 20 mg | Part 2 (MAD): ATH-399A 40 mg | Part 2 (MAD): ATH-399A 40 mg, Older
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 12 | 8 | 6 | 6 | 6
hours | 7 [2 to 12] | 8.009 [6 to 12] | 4.500 [2 to 8] | 4.059 [3 to 8.017] | 7 [3 to 8] | 6.009 [4 to 16] | 4 [2 to 12] | 5.009 [2 to 12] | 7 [4 to 8.017] | 8.017 [2 to 23.517]

17. Secondary Outcome: λz
Description: PK parameter: Individual Estimate Of The Terminal Elimination Rate Constant (λz) for Part 1a, Part 1b and Part 2. λz was calculated based on several PK blood sampling at times provided in the Outcome Measure Time Frame.
Time Frame: as for outcome 13
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | Part 1a (SAD): ATH-399A 5 mg | Part 1a (SAD): ATH-399A 10 mg | Part 1a (SAD): ATH-399A 20 mg | Part 1a (SAD): ATH-399A 40 mg | Part 1a (SAD): ATH-399A 80 mg | Part 1b (Food Effect): ATH-399A 40 mg, Fed | Part 1b (Food Effect): ATH-399A 40 mg, Fasted | Part 2 (MAD): ATH-399A 20 mg | Part 2 (MAD): ATH-399A 40 mg | Part 2 (MAD): ATH-399A 40 mg, Older
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 12 | 8 | 6 | 5 | 4
1/hr | 0.0304 (0.0081) | 0.0308 (0.0062) | 0.0363 (0.0069) | 0.0269 (0.0057) | 0.0250 (0.0041) | 0.0253 (0.0052) | 0.0261 (0.0047) | 0.0286 (0.0041) | 0.0264 (0.0026) | 0.0235 (0.0028)

18. Secondary Outcome: t½ el
Description: PK parameter: Terminal Elimination Half-Life (t½ el) for Part 1a, Part 1b and Part 2. T1/2 el was calculated based on several PK blood sampling at times provided in the Outcome Measure Time Frame.
Time Frame: as for outcome 13
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part 1a (SAD): ATH-399A 5 mg | Part 1a (SAD): ATH-399A 10 mg | Part 1a (SAD): ATH-399A 20 mg | Part 1a (SAD): ATH-399A 40 mg | Part 1a (SAD): ATH-399A 80 mg | Part 1b (Food Effect): ATH-399A 40 mg, Fed | Part 1b (Food Effect): ATH-399A 40 mg, Fasted | Part 2 (MAD): ATH-399A 20 mg | Part 2 (MAD): ATH-399A 40 mg | Part 2 (MAD): ATH-399A 40 mg, Older
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 12 | 8 | 6 | 5 | 4
hours | 23.86 (4.80) | 23.32 (4.96) | 19.71 (4.01) | 26.77 (5.59) | 28.31 (4.65) | 28.48 (5.62) | 27.32 (4.82) | 24.63 (3.28) | 26.44 (2.59) | 29.85 (3.44)

19. Secondary Outcome: Cmax, ss
Description: PK parameter: Maximal Observed Concentration at steady state (Cmax, ss) for Part 2. Cmax,ss was calculated based on several PK blood sampling at times provided in the Outcome Measure Time Frame.
Time Frame: Part 2 only: Day 12 Pre-dose (within 2 hours of dosing) and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours.
Population: Cmax ss has been analyzed only in patients included in Part 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 2 (MAD): ATH-399A 20 mg | Part 2 (MAD): ATH-399A 40 mg | Part 2 (MAD): ATH-399A 40 mg, Older
Number analyzed (Participants) | 6 | 5 | 4
ng/mL | 14.98 (6.89) | 51.88 (34.86) | 46.04 (21.52)

20. Secondary Outcome: Cmin ss
Description: PK parameter: Minimal Observed Concentration at steady-state (Cmin ss) for Part 2. Cmin was calculated based on several PK blood sampling at times provided in the Outcome Measure Time Frame.
Time Frame: as for outcome 19
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Part 2 (MAD): ATH-399A 40 mg2: Each participant received ATH-399A 40 mg once daily from Day 1 to Day 12. Participants underwent a supervised fast for at least 10 hours prior to dosing, followed by an additional 4 hours of fasting post-dose.
Arm/Group | Part 2 (MAD): ATH-399A 20 mg | Part 2 (MAD): ATH-399A 40 mg2 | Part 2 (MAD): ATH-399A 40 mg, Older
Number analyzed (Participants) | 6 | 5 | 4
ng/mL | 6.25 (2.16) | 17.91 (6.87) | 20.39 (6.89)

21. Secondary Outcome: Cavg
Description: PK parameter: Average Plasma Concentration (Cavg) for Part 2. Cavg was calculated based on several PK blood sampling at times provided in the Outcome Measure Time Frame.
Time Frame: as for outcome 19
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 40mg: Part 2 (MAD): ATH-399A 40mg
- 40 mg (older): Part 2 (MAD) ATH-399A 40 mg (older)
Arm/Group | Part 2 (MAD): ATH-399A 20 mg | 40mg | 40 mg (older)
Number analyzed (Participants) | 6 | 5 | 4
ng/mL | 10.47 (3.41) | 30.21 (14.42) | 32.28 (12.42)

22. Secondary Outcome: Tmax, ss
Description: PK parameter: Time When The Maximal Concentration Is Observed at Steady State (Tmax, ss) for Part 2. Tmax, ss was calculated based on several PK blood sampling at times provided in the Outcome Measure Time Frame.
Time Frame: as for outcome 19
Measure: Median (Full Range); unit: hours
Arm/Group | Part 2 (MAD): ATH-399A 20 mg | Part 2 (MAD): ATH-399A 40 mg | Part 2 (MAD): ATH-399A 40 mg, Older
Number analyzed (Participants) | 6 | 5 | 4
hours | 5 [4 to 8] | 4 [3 to 12] | 5.5 [1 to 24]

23. Secondary Outcome: AUC0-τ (AUC0-24 at Day 12 Dose) for Part 2
Description: PK parameter: Area Under The Concentration-Time Curve For One Dosing Interval (Τ) (AUC0-τ) [i.e., AUC0-24 on Day 12 dose] for Part 2 only. Value was calculated based on several PK blood sampling at times provided in the Outcome Measure Time Frame.
Time Frame: as for outcome 19
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 2 (MAD): ATH-399A 20 mg | Part 2 (MAD): ATH-399A 40 mg | Part 2 (MAD): ATH-399A 40 mg, Older
Number analyzed (Participants) | 6 | 5 | 4
h*ng/mL | 251.24 (81.96) | 725.06 (345.98) | 774.81 (298.05)

24. Secondary Outcome: AUC0-t on Day 1 Dose for Part 2
Description: PK parameter: Area Under The Concentration-Time Curve AUC0-t (i.e., AUC0-24 on Day 1 dose only) for Part 2
Time Frame: Part 2 only: Day 1 Pre-dose (within 2 hours of dosing) and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 2 (MAD): ATH-399A 20 mg | Part 2 (MAD): ATH-399A 40 mg | Part 2 (MAD): ATH-399A 40 mg, Older
Number analyzed (Participants) | 6 | 6 | 6
h*ng/mL | 83.99 (34.09) | 208.14 (126.00) | 186.80 (88.77)

25. Primary Outcome: Laboratory Parameter: Creatinine Value
Description: Laboratory parameter: Creatinine level on Day 1
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Part 1a (SAD): ATH-399A 5 mg | Part 1a (SAD): ATH-399A 10 mg | Part 1a (SAD): ATH-399A 20 mg | Part 1a (SAD): ATH-399A 40 mg | Part 1a (SAD): ATH-399A 80 mg | Part 1a (SAD): Placebo | Part 1b (Food Effect): ATH-399A 40 mg, Fed | Part 1b (Food Effect): ATH-399A 40 mg, Fasted | Part 2 (MAD): ATH-399A 20 mg | Part 2 (MAD): ATH-399A 40 mg | Part 2 (MAD): ATH-399A 40 mg, Older | Part 2 (MAD): Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 12 | 8 | 6 | 6 | 6 | 6
μmol/L | 79.2 (16.87) | 78.5 (19.95) | 64.8 (13.27) | 88.3 (8.02) | 70.2 (9.06) | 76.6 (10.86) | 76.5 (15.26) | 76.4 (16.37) | 87.5 (14.46) | 111.2 (15.43) | 84.0 (11.24) | 87.3 (14.96)

26. Primary Outcome: Laboratory Parameter: Glucose
Description: Laboratory parameter: Glucose level measured on Day 1
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part 1a (SAD): ATH-399A 5 mg | Part 1a (SAD): ATH-399A 10 mg | Part 1a (SAD): ATH-399A 20 mg | Part 1a (SAD): ATH-399A 40 mg | Part 1a (SAD): ATH-399A 80 mg | Part 1a (SAD): Placebo | Part 1b (Food Effect): ATH-399A 40 mg, Fed | Part 1b (Food Effect): ATH-399A 40 mg, Fasted | Part 2 (MAD): ATH-399A 20 mg | Part 2 (MAD): ATH-399A 40 mg | Part 2 (MAD): ATH-399A 40 mg, Older | Part 2 (MAD): Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 12 | 8 | 6 | 6 | 6 | 6
mmol/L | 4.35 (0.797) | 4.07 (0.585) | 4.16 (0.657) | 4.62 (0.983) | 4.23 (0.779) | 4.04 (0.782) | 4.95 (0.894) | 4.84 (0.907) | 4.43 (0.441) | 4.43 (0.568) | 3.85 (0.356) | 4.58 (0.313)

ADVERSE EVENTS:
Time Frame: Continuously during study period from baseline to follow-up visit: Part 1a: Day-1 to Day 8, Part 1b: Day-1 to Day 16; and Part 2: Day -1 to Day 19
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study drug, whether or not considered related to the study drug.
Arm/Group | Part 1a (SAD): ATH-399A 5 mg | Part 1a (SAD): ATH-399A 10 mg | Part 1a (SAD): ATH-399A 20 mg | Part 1a (SAD): ATH-399A 40 mg | Part 1a (SAD): ATH-399A 80 mg | Part 1a (SAD): Placebo | Part 1b (Food Effect): ATH-399A 40 mg, Fed | Part 1b (Food Effect): ATH-399A 40 mg, Fasted | Part 2 (MAD): ATH-399A 20 mg | Part 2 (MAD): ATH-399A 40 mg | Part 2 (MAD): ATH-399A 40 mg, Older | Part 2 (MAD): Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10 | 0/12 | 0/8 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10 | 0/12 | 0/8 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/6 | 1/6 | 1/6 | 2/6 | 1/6 | 2/10 | 3/12 | 1/8 | 3/6 | 2/6 | 3/6 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1a (SAD): ATH-399A 5 mg (N=6) | Part 1a (SAD): ATH-399A 10 mg (N=6) | Part 1a (SAD): ATH-399A 20 mg (N=6) | Part 1a (SAD): ATH-399A 40 mg (N=6) | Part 1a (SAD): ATH-399A 80 mg (N=6) | Part 1a (SAD): Placebo (N=10) | Part 1b (Food Effect): ATH-399A 40 mg, Fed (N=12) | Part 1b (Food Effect): ATH-399A 40 mg, Fasted (N=8) | Part 2 (MAD): ATH-399A 20 mg (N=6) | Part 2 (MAD): ATH-399A 40 mg (N=6) | Part 2 (MAD): ATH-399A 40 mg, Older (N=6) | Part 2 (MAD): Placebo (N=6)
COVID-19, conjunctivitis, asymptomatic bacteriuria, nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasal congestion, nasal dryness, oropharyngeal pain, hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure decreased, blood pressure increased, blood creatine phosphokinase increased, electroc (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Accelerated idioventricular rhythm, ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal sensation in eye, conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry mouth, abdominal discomfort, constipation, abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope, headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain, musculoskeletal chest pain, neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2024-09-26): https://cdn.clinicaltrials.gov/large-docs/84/NCT06088784/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/84/NCT06088784/SAP_001.pdf